CLINICAL TRIAL: NCT01298284
Title: Endoscopic Treatment Alone Versus Combined Propranolol and Endoscopic Treatment of Acute Variceal Hemorrhage in Patients With HCC:a Randomized Trial
Brief Title: A Trial of EVL\GVS Alone vs. EVL\GVS Combined Propranolol
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: MING CHIH HOU,M.D / Taipei Veterans General Hospital,Taiwan, Taipei Veterans General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: V99C1-026; IRB:98-09-09 (Other: IRB:98-09-09)
Record Dates: First submitted 2010-10-04; First posted 2011-02-17 (Estimated); Last update posted 2011-06-15 (Estimated); Status verified 2011-06

CONDITIONS: Liver Cirrhosis; Hepatoma
Keywords: Variceal bleeding; portal hypertension; hepatocelluar carcinoma; endoscopic variceal ligation; non-selective beta-blocker; rebleeding
MeSH Terms: conditions — Liver Cirrhosis; Carcinoma, Hepatocellular; Hypertension, Portal | interventions — Propranolol

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- EVL\GVS Alone (No Intervention): Endoscopic ligation treatment in the 2nd prevention of gastroesophageal variceal bleeding in patients with HCC
- EVL\GVS Combined Propranolol (Active Comparator): Propranolol and endoscopic ligation treatment is used for 2nd prevention of gastroesophageal variceal bleeding in patients with HCC.
  <EVL\GVS Combined Propranolol>
  Interventions: Drug: propranolol

INTERVENTIONS:
Drug: propranolol — Starting from 20 mg daily, titrated weekly to decrease heart rate more than 25 % of baseline, administrated during the whole study period
  Other Names: Inderal,Cardolol
  Arms: EVL\GVS Combined Propranolol

SUMMARY:
New strategy to improve the outcomes in patients with HCC and acute variceal bleeding. NSBB added to endoscopic ligation may further reduce rebleeding in cirrhotic patients.

DETAILED DESCRIPTION:
Gastroesophageal vaiceal bleeding is a major complication of portal hypertension. Gastroesophageal variceal bleeding is characteristic of high rebleeding rate and mortality. Thanks to the recent advance of treatment including immediate vasoactive agents (such as somatostatin and vasopressin analogue for acute bleeding), non-selective beta-blocker (NSBB) for prevention of bleeding, prophylactic antibiotics, endoscopic variceal ligation, endoscopic cyanoacrylate injection , combination treatment and general improvement of care for patients with acute variceal bleeding, the rebleeding rate and mortality has a marked reduction. However, hepatocellular carcinoma (HCC) is a distinct group characteristic of very poor prognosis in patients in portal hypertensive patients when compared to those of liver cirrhosis only. Therefore it needs to specially clarify their treatment strategy, particularly in Taiwan, a highly prevalent area of HCC.

In patients of HCC presenting acute variceal bleeding, the rebleeding is around 50% doubled that of patients with cirrhosis only and bleeding mortality also more than 50%. The trend is not changed even after introduction of immediate use of vasoactive agents and endoscopic ligation. The poor outcome is because that HCC patients usually have arterioporal shunting or portal vein thrombosis and higher portal pressure. Moreover, their liver function deteriorated faster. Both high portal pressure and poor liver function are major determinant of hemostatic outcomes. Therefore, it is important to find a new strategy to improve the outcomes in patients with HCC and acute variceal bleeding.NSBB added to endoscopic ligation may further reduce rebleeding in cirrhotic patients. However, whether the hypotensive effect of NSBB is adequate to prevent rebleeding in patients with HCC who usually has higher portal pressure in not known. In addition, concomitant rapid deterioration of liver function might also dampen NSBB effects. Furthermore, due to faster deterioration of general condition, the tolerance of NSBB in these patients might be remarkable and lead to a higher withdrawal rate. Therefore, it is very important to clarify whether there is additive therapeutic effect of NSBB to endoscopic treatment in the 2nd prevention of gastroesophageal variceal bleeding in patients with HCC.

Therefore, the investigators design a study to randomize patients with HCC and acute variceal bleeding to endoscopic treatment alone and combination with endoscopic treatment and NSBB. This is the two years study.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of HCC, endoscopically proven gastroesophageal variceal bleeding
* Aged 18 to 80

Exclusion Criteria:

* Had a terminal illness of any major organ system,such as heart failure, kidney failure, COPD

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2009-10; Primary Completion 2010-06 (Actual); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Rebleeding | 1 years

SECONDARY OUTCOMES:
complication surivial | 1 years

CONTACTS AND LOCATIONS:
Overall Officials: Ming-Chih Hou, MD, Principal Investigator — Taipei Veterans General Hospital, Taiwan
Locations (1):
- Veteran General Hospital-Taipei, Taipei, Taiwan, Taiwan